CLINICAL TRIAL: NCT04249765
Title: Hand Strength And Hand-Reaction Parameters Of Post Millennial: An Example Of Students' Group In Central Anatolia
Acronym: HS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Collaborators: Atılım University (Other)
Responsible Party: Principal Investigator, İSMAİL CEYLAN, Head of Hand Therapy Clinic, Ahi Evran University Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 12068451748
Record Dates: First submitted 2020-01-26; First posted 2020-01-31 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hand Grasp
Keywords: Hand function

STUDY DESIGN:
Intervention Model Description: Cross sectional research design with data collected over one semester.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hand strength (Experimental): Grip Strength The participants sat upright on a chair with their feet supported. The tested arm was positioned on a table with the shoulders slightly abducted and neutrally rotated, the elbow in 90° of flexion, the forearm in 0° between pronation and supination, and the wrist in neutral resting position. The participants were instructed to maintain that position during the test. The grip strength of both hands was measured using the Hand Dynamometer
  3. Pinch Strength Participants were seated at a table on which the dynamometers were positioned.
  The subjects were told to keep their elbow flexed without resting their arm or the grip handle of the dynamometer.
  Interventions: Other: Assessing grasping force, pinch force,

INTERVENTIONS:
Other: Assessing grasping force, pinch force, — Grip Strength The participants sat upright on a chair with their feet supported. The tested arm was positioned on a table with the shoulders slightly abducted and neutrally rotated, the elbow in 90° of flexion, the forearm in 0° between pronation and supination, and the wrist in neutral resting position. The participants were instructed to maintain that position during the test. The grip strength of both hands was measured using the Hand Dynamometer.
  3. Pinch Strength Participants were seated at a table on which the dynamometers were positioned. The subjects were told to keep their elbow flexed without resting their arm or the grip handle of the dynamometer on the table.

SUMMARY:
The aim of this research is to find out whether there exists a correlation between such important characteristic of individual's hand performance as grip strength, pinch strength, and the hand reaction. In addition, it will be investigated whether there is a change in normative values of this age group in relation to modern lifestyle. The study includes statistical data analysis and interpretation of the derived outcomes.

DETAILED DESCRIPTION:
Objective: To investigate correlation between grip force, pinch strength and hand reaction in a group of post-millennial in Central Anatolia, and also to provide a comparison to previously available results on millennial.

Methods: Experimental data were collected by healthy subjects, who are university students. The sample comprises females and males, consented to participate in the study. The ages of the subjects will range from 18 to 25 years. Grip strength will measure with hand dynamometer and pinch strength will measure with pinch meter. Hand reaction will test with the Ruler Drop Test.

For each subject, body mass, height and hand preference will be record. The study will be completed in accordance with the norms of the Declaration of Helsinki and was approved by the ethics committee of the University of Atilim (Turkey).

The collected data will be undergone statistical analysis to extract any feasible conclusions. First, the correlation coefficients will be found to determine whether there is a noticable relationship between the independent variables grip strength and pinch strength versus the dependent variable ruler drop test. The calculated sample correlation coefficients have been tested for the significance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* History of any upper extremity pain or injury

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2021-03-25 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | Measurements will assessed in 1 month and data will analysed in 2 months.
  The participants will sit upright on a chair with their feet supported. The tested arm will positioned on a table with the shoulders slightly abducted and neutrally rotated, the elbow in 90° of flexion, the forearm in 0° between pronation and supination, and the wrist in neutral resting position. The grip strength of both hands will measured using the Hand Dynamometer. Results will be evaluated in kilograms.

SECONDARY OUTCOMES:
Hand Pinch Strength | Measurements will assessed in 1 month and data will analysed in 2 months.
  Participants were seated at a table on which the dynamometers were positioned. The subjects were told to keep their elbow flexed without resting their arm or the grip handle of the dynamometer on the table. Results will be evaluated in kilograms.
Ruler Drop Test | Measurements will assessed in 1 month and data will analysed in 2 months.
  During the test, the students had to sit having the upper arm forming an angle of 90 degrees with the mid forearm, which lies on a flat horizontal table surface. The hand is required to be open and positioned at the edge of the surface. Results will be evaluated in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Turan, Doç. Dr., Study Director — Atılım University
Locations (1):
- Atılım University, Ankara, Middle Anatolia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No